CLINICAL TRIAL: NCT01620918
Title: Soft Tissue Responses Around Nanostructured Calcium-phosphate-coated Implant Abutments on Dental Implants: Histological, Genetic and Clinical Evaluation in Smokers and Non-smokers.
Acronym: STRANDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012/341
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2021-12-01 (Actual); Status verified 2021-11

CONDITIONS: Missing Several Teeth; Minimum of 2 Dental Implants Needed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 2 types of healing abutment (Experimental): Patients who are in need of minimal 2 dental implants, who will receive both types of healing abutments.
  Interventions: Procedure: normal healing abutment; Procedure: nano-structured healing abutment

INTERVENTIONS:
Procedure: normal healing abutment — Patient receives the normal, uncoated healing abutment on 1 of his (minimal 2) dental implants.
Procedure: nano-structured healing abutment — Patient receives the nano-structured healing abutment on 1 of his (minimal 2) dental implants.

SUMMARY:
* Baseline:

  * Standard preparation of the osteotomy
  * Placement of 2 dental implants
  * On each implant one of both types of healing abutments is placed
  * Suturing
  * Standardized radiography to measure bone-levels at baseline
  * Digital impression of the surrounding gingiva with an intra-oral scanner (a non-invasive method) to measure the baseline level of the gingiva
* 2 weeks after Baseline:

  o Removal of the sutures
* 4 weeks after Baseline:

  * A 2nd digital impression of the soft tissue with an intra-oral scanner
  * Collecting crevicular fluid by placing paperpoints in the provided apertures in the healing abutments for 60 seconds without bleeding.
  * Measuring of the pocket depth in the provided apertures in the healing abutments with an automated probe.
  * Removal of the Healing Abutment with the attached soft tissue en-bloque.
  * Placement of a new, regular, Encode Healing Abutment.
* 10 weeks after Baseline:

  * Start of standard prosthetic procedure. In this study we expect that the soft tissue attachment (i.e. the gingival attachment) will be stronger and earlier achieved at the nano-structured healing abutments than at the normal, uncoated healing abutments. This would lead to a more stable soft tissue complex on the long rung and thus providing a more predictable aesthetic outcome. Secondly, a stronger attachment would mean a stronger barrier against micro-organisms and might influence the occurrence of peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for this study if they are in need of minimum 2 dental implants and have sufficient bone to place these implants

Exclusion Criteria:

* All patients with limited bone
* Periodontally compromised patients
* Patients who took antibiotics 3 months before implantation
* Patients with uncontrolled diabetes
* Pregnant patients
* Patients who received radiotherapy in the head/neck region
* Patients under chemotherapy
* Patients who had intravenous use of bisphosphonates

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The soft-tissue attachment around 2 different surfaces at 4 weeks post-implantation. | at 4 weeks post-implantation
  Genetic evaluation (through Polymerase Chain Reaction, PCR, the tissue will be detected for certain growth factors), histomorphometric analysis to measure the actual percentage of the surface on which the gingiva is attached to, clinical evaluation of the strength of the attachment through means of an automated probe.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo De Bruyn, DDS, MSc, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium